CLINICAL TRIAL: NCT03448588
Title: Effect of Selenium Deficiency on Thyroid Function
Brief Title: Research on Association Between Selenium Deficiencies and Change of Thyroid Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liuyanping, Dietitian, Peking Union Medical College Hospital
Other Study IDs: Liuyanping3
Record Dates: First submitted 2018-02-07; First posted 2018-02-28 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Selenium Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group with normal T4 level or T4/T3: participants with T4 within 4.3-12.5ug/dl and ratio of T4/T3(T4(ug/dl)/T3 (ng/ml)) ≤7.52, which are considered to be normal T4 level and T4/T3.
  Interventions: Diagnostic Test: detection of serum selenium
- group with elevated T4 level or T4/T3: participants with T4 more than 12.5ug/dl and ratio of T4/T3(T4(ug/dl)/T3 (ng/ml)) > 7.52, which are considered to be elevated T4 level and T4/T3.
  Interventions: Diagnostic Test: detection of serum selenium

INTERVENTIONS:
Diagnostic Test: detection of serum selenium — For this case-control study, no intervention will be administered to participants, only serum sample will be collected for selenium assessment

SUMMARY:
As one of the essential micronutrients, selenium has important biological functions. However, an effective and convenient method for evaluation of selenium nutritional status has not yet been established. Previous literature has disclosed effect of selenium deficiency on inactivating glutathion peroxidase and deiodinase, which may cause decreased conversion from thyroxine ( T4) to triiodothyronine (T3). A case-control study is designed to demonstrate the association between selenium deficiency and abnormally elevated T4 or T4/T3, which may provide more clues for establishing effective selenium assesment methods.

ELIGIBILITY:
Inclusion Criteria:

* with normal free triiodothyronine( FT3), free thyroxine (FT4) and thyroid-stimulating hormone (TSH).
* without thyroid hormone replacement therapy
* without medical history of thyroid surgery
* without iodine radiotherapy;

Exclusion Criteria:

* acute critical illness in the latest 1 year;
* weight fluctuation by more than 5% in the latest 3 months;
* eating disorders
* neuropsychological disorders
* allergy to corn or yeast
* fail to give informed consents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from volunteers who undergo health examination in Peking Union Medical College Hospital and meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
between-group difference in serum selenium | up to 24 weeks
  comparison of the mean serum selenium between the two groups

SECONDARY OUTCOMES:
between-group difference in serum deiodinase activity | up to 24 weeks
  comparison of the mean deiodinase activity between the two groups
between-group difference in erythrocyte glutathione peroxidase activity | up to 24 weeks
  comparison of the mean erythrocyte glutathione peroxidase activity between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No